CLINICAL TRIAL: NCT03619512
Title: Genomic and Proteomic Study of Richter Syndrome
Brief Title: Genomic and Proteomic Study of Richter Syndrome (CGPSR)
Acronym: CGPSR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: French Innovative Leukemia Organization (FILO) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-A01978-45; PSS2017/CGPSR-BROSÉUS/VS (Other: CHRU Nancy)
Record Dates: First submitted 2018-07-19; First posted 2018-08-08 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Richter Syndrome
Keywords: Richter Syndrome; Genomics; Proteomics; Chemotherapy resistance
MeSH Terms: interventions — Exome Sequencing; Sequence Analysis, RNA; Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Richter Syndrom at diagnosis: patients diagnosed with Richter Syndrom, for whom a suitable lymph node biopsy at diagnosis is available.
  Interventions: Genetic: Whole exome sequencing.; Genetic: RNA sequencing; Other: Mass spectrometry
- Primitive Diffuse Large B-Cell Lymphoma: patients diagnosed with a primitive Large B-Cell Lymphoma, for whom a suitable lymph node biopsy at diagnosis is available.
  Interventions: Genetic: Whole exome sequencing.; Genetic: RNA sequencing; Other: Mass spectrometry
- Other secundary Diffuse Large B-Cell Lymphoma: patients diagnosed with a secundary Large B-Cell Lymphoma (different from Richter Syndrom), for whom a suitable lymph node biopsy at diagnosis is available.
  Interventions: Genetic: Whole exome sequencing.; Genetic: RNA sequencing; Other: Mass spectrometry
- Control group with no tumor involvment of lymph nodes: patients for whom a diagnostic lymph node biopsy has been performed, which did not conclude to any tumoral lymph node involvment.
  Interventions: Genetic: Whole exome sequencing.; Genetic: RNA sequencing; Other: Mass spectrometry

INTERVENTIONS:
Genetic: Whole exome sequencing. — Retrospective biological exploration of the samples, including tumoral DNA exploration.
Genetic: RNA sequencing — Characterization of tumor transcriptomic profile.
Other: Mass spectrometry — Characterization of tumor proteomic profiles.

SUMMARY:
Biological study on Richter Syndrome (RS), an agressive lymphoma that arises from Chronic Lymphocytice Leukemia (CLL). RS presents with the same histological aspect as primitive Diffuse Large B-Cell Lymphoma (DLBCL), but is associated with a poor prognosis, due to chemorefractoriness.

This study aims at understanding the biological determinants of chemotherapy resistance in Richter Syndrome.

DETAILED DESCRIPTION:
With the help of the French National Research Group on CLL (FILO / French Innovative Leukemia Organization), the investigators are currently gathering fresh frozen cell pellets at CLL stage, and lymph node biopsies at Richter stage. The investigators also gathered lymph node biopsies from DLBCL, as a reference group.

The investigators will perform genomic and proteomic comparative studies between CLL and Richter, as well as between Richter and primitive DLBCL, to understand the biological determinants of clonal evolution and chemorefractoriness of Richter Syndrom.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a Diffuse Large B-Cell Lymphoma arising in the context of a Chronic Lymphocytic Leukemia (group 1) or diagnosis of a primitive Diffuse Large B-Cell Lymphoma (group 2), or diagnosis of a Diffuse Large B-Cell Lymphoma arising in a context of small cells lymphoma, excluding CLL (group 3), or benefit from a diagnostic lymph node biopsy that did not reveal any tumor involvment (primitive or metastatic) (group 4).
* Patients must benefit from a lymph node biopsy at diagnosis.
* Patients must be followed by a FILO (French Innovative Leukemia Organization) member
* Histology of Diffuse Large B-Cell Lymphoma or Hodgkin histology.
* Suitable clinical data available.
* Samples must meet the following requirement :RIN (RNA Integrity Number) > 5 et DIN (DNA Integrity Number) > 6.5.

Exclusion Criteria:

• Samples that do not meet the inclusion criteria (insufficient clinical data, analysis impossible due to insufficient sample quality).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Diagnosis of Diffuse Large B-Cell Lymphoma arising in the context of a Chronic Lymphocytic Leukemia (group 1).
  * Diagnosis of Diffuse Large B-Cell Lymphoma de novo (group 2).
  * Diagnosis of Diffuse Large B-Cell Lymphoma arising in a context of small cells lymphoma, excluding CLL (group 3).
  * Patients who benefited from a diagnostic lymph node biopsy that did not reveal any tumor involvment (primitive or metastatic) (group 4).
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-09-05 (Estimated)

PRIMARY OUTCOMES:
Whole exome sequencing data using next generation sequencing method | 3 years
  Comparison between the DNA sequences from Richter syndrome samples and DNA sequences from primitive DLBCL samples to identify a set of mutations that are specific to Richter syndrome.
  For each position, the result is "mutated" or "unmutated".
RNA sequencing data using next generation sequencing method | 3 years
  Measurment of gene expression for all genes. Comparison of these expression levels between Richter samples, primitive DLBCL samples and normal lymph nodes to identifiy a set of genes which expression levels are different in Richter samples compared primitive DLBCL and normal lymph nodes.
  Gene expression is a quatitative value. This set of genes forms a specific "transcriptomic signature" of Richter syndrome.
Proteomic analysis using mass spectrometry | 3 years
  Mass spectrometry allows identification and measurment of the expression level of the 5,000 most expressed proteins in a sample. The investigators want to compare the protein expression levels between Richter samples, primitive DLBCL samples and normal lymph nodes to identifiy a set of proteins that are highly expressed in Richter samples (but not in primitive DLBCL or normal lymph nodes). This set of proteins forms a specific "proteomic signature" of Richter.
  Protein expression is a quatitative value expressed as an absolute number of copies in a cell.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Broseus, MD, PhD, Principal Investigator — Central Hospital, Nancy, France; Pierre Feugier, MD, PhD, Study Director — Central Hospital, Nancy, France
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi D, Spina V, Forconi F, Capello D, Fangazio M, Rasi S, Martini M, Gattei V, Ramponi A, Larocca LM, Bertoni F, Gaidano G. Molecular history of Richter syndrome: origin from a cell already present at the time of chronic lymphocytic leukemia diagnosis. Int J Cancer. 2012 Jun 15;130(12):3006-10. doi: 10.1002/ijc.26322. Epub 2011 Aug 25. PMID 21796624
- [Background] Ferreira PG, Jares P, Rico D, Gomez-Lopez G, Martinez-Trillos A, Villamor N, Ecker S, Gonzalez-Perez A, Knowles DG, Monlong J, Johnson R, Quesada V, Djebali S, Papasaikas P, Lopez-Guerra M, Colomer D, Royo C, Cazorla M, Pinyol M, Clot G, Aymerich M, Rozman M, Kulis M, Tamborero D, Gouin A, Blanc J, Gut M, Gut I, Puente XS, Pisano DG, Martin-Subero JI, Lopez-Bigas N, Lopez-Guillermo A, Valencia A, Lopez-Otin C, Campo E, Guigo R. Transcriptome characterization by RNA sequencing identifies a major molecular and clinical subdivision in chronic lymphocytic leukemia. Genome Res. 2014 Feb;24(2):212-26. doi: 10.1101/gr.152132.112. Epub 2013 Nov 21. PMID 24265505
- [Result] Rossi D, Cerri M, Capello D, Deambrogi C, Rossi FM, Zucchetto A, De Paoli L, Cresta S, Rasi S, Spina V, Franceschetti S, Lunghi M, Vendramin C, Bomben R, Ramponi A, Monga G, Conconi A, Magnani C, Gattei V, Gaidano G. Biological and clinical risk factors of chronic lymphocytic leukaemia transformation to Richter syndrome. Br J Haematol. 2008 Jun;142(2):202-15. doi: 10.1111/j.1365-2141.2008.07166.x. Epub 2008 May 19. PMID 18492108
- [Result] Parikh SA, Rabe KG, Call TG, Zent CS, Habermann TM, Ding W, Leis JF, Schwager SM, Hanson CA, Macon WR, Kay NE, Slager SL, Shanafelt TD. Diffuse large B-cell lymphoma (Richter syndrome) in patients with chronic lymphocytic leukaemia (CLL): a cohort study of newly diagnosed patients. Br J Haematol. 2013 Sep;162(6):774-82. doi: 10.1111/bjh.12458. Epub 2013 Jul 11. PMID 23841899
- [Result] Rossi D, Spina V, Deambrogi C, Rasi S, Laurenti L, Stamatopoulos K, Arcaini L, Lucioni M, Rocque GB, Xu-Monette ZY, Visco C, Chang J, Chigrinova E, Forconi F, Marasca R, Besson C, Papadaki T, Paulli M, Larocca LM, Pileri SA, Gattei V, Bertoni F, Foa R, Young KH, Gaidano G. The genetics of Richter syndrome reveals disease heterogeneity and predicts survival after transformation. Blood. 2011 Mar 24;117(12):3391-401. doi: 10.1182/blood-2010-09-302174. Epub 2011 Jan 25. PMID 21266718
- [Result] Fangazio M, De Paoli L, Rossi D, Gaidano G. Predictive markers and driving factors behind Richter syndrome development. Expert Rev Anticancer Ther. 2011 Mar;11(3):433-42. doi: 10.1586/era.10.237. PMID 21417856
- [Result] Rossi D, Rasi S, Spina V, Fangazio M, Monti S, Greco M, Ciardullo C, Fama R, Cresta S, Bruscaggin A, Laurenti L, Martini M, Musto P, Forconi F, Marasca R, Larocca LM, Foa R, Gaidano G. Different impact of NOTCH1 and SF3B1 mutations on the risk of chronic lymphocytic leukemia transformation to Richter syndrome. Br J Haematol. 2012 Aug;158(3):426-9. doi: 10.1111/j.1365-2141.2012.09155.x. Epub 2012 May 10. No abstract available. PMID 22571487
- [Result] Fabbri G, Rasi S, Rossi D, Trifonov V, Khiabanian H, Ma J, Grunn A, Fangazio M, Capello D, Monti S, Cresta S, Gargiulo E, Forconi F, Guarini A, Arcaini L, Paulli M, Laurenti L, Larocca LM, Marasca R, Gattei V, Oscier D, Bertoni F, Mullighan CG, Foa R, Pasqualucci L, Rabadan R, Dalla-Favera R, Gaidano G. Analysis of the chronic lymphocytic leukemia coding genome: role of NOTCH1 mutational activation. J Exp Med. 2011 Jul 4;208(7):1389-401. doi: 10.1084/jem.20110921. Epub 2011 Jun 13. PMID 21670202
- [Result] Chigrinova E, Rinaldi A, Kwee I, Rossi D, Rancoita PM, Strefford JC, Oscier D, Stamatopoulos K, Papadaki T, Berger F, Young KH, Murray F, Rosenquist R, Greiner TC, Chan WC, Orlandi EM, Lucioni M, Marasca R, Inghirami G, Ladetto M, Forconi F, Cogliatti S, Votavova H, Swerdlow SH, Stilgenbauer S, Piris MA, Matolcsy A, Spagnolo D, Nikitin E, Zamo A, Gattei V, Bhagat G, Ott G, Zucca E, Gaidano G, Bertoni F. Two main genetic pathways lead to the transformation of chronic lymphocytic leukemia to Richter syndrome. Blood. 2013 Oct 10;122(15):2673-82. doi: 10.1182/blood-2013-03-489518. Epub 2013 Sep 4. PMID 24004666
- [Result] Scandurra M, Rossi D, Deambrogi C, Rancoita PM, Chigrinova E, Mian M, Cerri M, Rasi S, Sozzi E, Forconi F, Ponzoni M, Moreno SM, Piris MA, Inghirami G, Zucca E, Gattei V, Rinaldi A, Kwee I, Gaidano G, Bertoni F. Genomic profiling of Richter's syndrome: recurrent lesions and differences with de novo diffuse large B-cell lymphomas. Hematol Oncol. 2010 Jun;28(2):62-7. doi: 10.1002/hon.932. PMID 20014148
- [Result] Fabbri G, Khiabanian H, Holmes AB, Wang J, Messina M, Mullighan CG, Pasqualucci L, Rabadan R, Dalla-Favera R. Genetic lesions associated with chronic lymphocytic leukemia transformation to Richter syndrome. J Exp Med. 2013 Oct 21;210(11):2273-88. doi: 10.1084/jem.20131448. Epub 2013 Oct 14. PMID 24127483
- [Result] Alizadeh AA, Eisen MB, Davis RE, Ma C, Lossos IS, Rosenwald A, Boldrick JC, Sabet H, Tran T, Yu X, Powell JI, Yang L, Marti GE, Moore T, Hudson J Jr, Lu L, Lewis DB, Tibshirani R, Sherlock G, Chan WC, Greiner TC, Weisenburger DD, Armitage JO, Warnke R, Levy R, Wilson W, Grever MR, Byrd JC, Botstein D, Brown PO, Staudt LM. Distinct types of diffuse large B-cell lymphoma identified by gene expression profiling. Nature. 2000 Feb 3;403(6769):503-11. doi: 10.1038/35000501. PMID 10676951
- [Derived] Moulin C, Guillemin F, Remen T, Bouclet F, Hergalant S, Quinquenel A, Dartigeas C, Tausch E, Lazarian G, Blanchet O, Lomazzi S, Chapiro E, Schneider C, Nguyen-Khac F, Davi F, Hunault M, Tomowiak C, Roos-Weil D, Siebert R, Thieblemont C, Cymbalista F, Laribi K, Bene MC, Stilgenbauer S, Guieze R, Feugier P, Broseus J. Clinical, biological, and molecular genetic features of Richter syndrome and prognostic significance: A study of the French Innovative Leukemia Organization. Am J Hematol. 2021 Sep 1;96(9):E311-E314. doi: 10.1002/ajh.26239. Epub 2021 Jun 2. No abstract available. PMID 34000073